CLINICAL TRIAL: NCT07042035
Title: Pharmacokinetic Study, Effectiveness, and Safety of the Tacrolimus Formulation Based on Melt-Dose® Technology (LCPT) as an Immunosuppressive Treatment for Lung Transplant Patients, Under Usual Clinical Practice Conditions.
Brief Title: Study of Tacrolimus Melt-Dose® for Lung Transplant Patients
Acronym: ESENCIAL
Status: Recruiting | Type: Observational
Sponsor: Chiesi España, S.A.U. (Other)
Collaborators: Trialance SCCL (Industry)
Responsible Party: Sponsor
Other Study IDs: CHI-TAC-2024-01
Record Dates: First submitted 2025-04-30; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lung Trasplant; Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate, under usual clinical practice conditions and with a 12-month follow-up , the most relevant pharmacokinetic parameters of tacrolimus metabolism and safety, in patients with recent lung transplant (unilateral or bilateral) treated with LCPT.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Patients who have received a first unilateral or bilateral lung transplant.
* Patients who have started oral treatment with tacrolimus using the LCPT formulation, with a once-daily dosage within the first 3 months post-transplant.
* Patients with a treatment duration expected to be ≥12 months.
* The patient (or their representative) can sign the informed consent to participate in the study.

Exclusion Criteria:

* Patients who have received a multi-organ transplant or have a history of any organ transplant, including lung.
* Patients with an estimated survival of <12 months
* Patients diagnosed with cystic fibrosis
* Patients diagnosed with scleroderma.
* Patients diagnosed with a systemic disease affecting the digestive system.
* Patients in any situation or condition that, in the investigator's opinion, makes participation inadvisable, such as any treatment that may interfere with the study.
* Patients who are participating or have participated in an interventional research study within 30 days prior to inclusion.
* Pregnant women, those planning to become pregnant, or those who are breastfeeding.
* Patients who are unable to complete the study.
* Patients who have not signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients after a first unilateral or bilateral lung transplant start treatment with rapid-release tacrolimus every 12 hours (IR-Tac formulation) and, after achieving a stable dose and before 3 months, switch to once-daily LCPT tacrolimus. These treatments will have been prescribed by the investigator following usual clinical practice, with no relation to inclusion in this study.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the most relevant pharmacokinetic parameters of tacrolimus metabolism and their relationship with clinical effectiveness and safety . | 1 year of follow up
  Cmin Tacrolimus dose

SECONDARY OUTCOMES:
To assess the pharmacokinetic parameters of LCPT ( concentration/dose ratio (C/D)). | 1 year
  Tacrolimus Cmin Tacrolimus dose Inter-patient tacrolimus variability. multiple measurements will be aggregated
To assess clinical effectiveness (acute rejection). | 1 year
  multiple measurements will be aggregated: Humoral rejection (circulating antibodies: number of patients and number of episodes) Acute clinical rejection (ACR); number of patients and number of episodesChronic Lung Allograft Dysfunction (CLAD); number of patients.
To assess lung function (spirometry). | 1 year
  Spirometry: Forced Vital Capacity (FVC) ml, percent of Forced Expiratory Volume in the first second (FEV1), and FEV1/FVC ratio.
To assess renal function (glomerular flow rate). | 1 year
  glomerular and flow rate
To assess the most frequent complications in lung transplant. | 1 year
  Assessment of immune activity indicators Patients with de novo Donor-Specific Antibody (dnDSA) detected after transplant - has or does not have (yes or no).
To assess adverse events. | 1 year
  Adverse Events (AEs), Adverse Drug Reactions (ADRs). AEs of special interest [assessed in case report form (CRF) on a case-by-case basis]: thrombotic microangiopathy (incidence after transplant); Reversible posterior encephalopathy (incidence after transplant); Pulmonary thromboembolism.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Chiesi España, Torre Realia BCN Plaza Europa 41-43, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No